CLINICAL TRIAL: NCT02534363
Title: Neurocognitive Effectiveness in Treatment of First-episode Non-affective Psychosis: a Randomized Comparison of Aripiprazole, Quetiapine and Ziprasidone Over 1 Year
Brief Title: Neurocognitive Effectiveness in Treatment of First-episode Non-affective Psychosis: 1-year Follow-up
Acronym: PAFIP2_nc1Y
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZQ2005_nc1Y; CI 2005-0308007 (Other Grant/Funding Number: SENY Fundació Research Grant CI 2005-0308007)
Record Dates: First submitted 2015-08-24; First posted 2015-08-27 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Cognition; Psychosis; Antipsychotic Agents; Treatment; Effectiveness; Aripiprazole; Quetiapine; Ziprasidone; Neurocognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aripiprazole & cognitive battery (Active Comparator): Aripiprazole 5-30 mg/day. Cognitive battery at baseline and at 1 year.
  Interventions: Drug: Aripiprazole; Behavioral: Cognitive battery
- Quetiapine & cognitive battery (Active Comparator): Quetiapine 100-600 mg/day. Cognitive battery at baseline and at 1 year.
  Interventions: Drug: Quetiapine; Behavioral: Cognitive battery
- Ziprasidone & cognitive battery (Active Comparator): Ziprasidone 40-160 mg/day. Cognitive battery at baseline and at 1 year.
  Interventions: Drug: Ziprasidone; Behavioral: Cognitive battery

INTERVENTIONS:
Drug: Aripiprazole — Oral, dose range 5-30 mg/day, once or twice a day, during study duration
  Other Names: Abilify
  Arms: Aripiprazole & cognitive battery
Drug: Quetiapine — Oral, dose range 100-600 mg/day, once or twice a day, during study duration
  Other Names: Seroquel
  Arms: Quetiapine & cognitive battery
Drug: Ziprasidone — Oral, dose range 40-160 mg/day, once or twice a day, during study duration
  Other Names: Zeldox
  Arms: Ziprasidone & cognitive battery
Behavioral: Cognitive battery — Completed in the following standardized sequence: 1-the Rey Auditory Verbal Learning Test (RAVLT); 2-WAIS-III digit symbol subtest; 3-Grooved Pegboard Test; 4-The Zoo Map Test; 5-Tower of London Test (ToL); 6-Rey Complex Figure (RCF); 7-Trail Making Test (TMT); 8-WAIS-III digits forward and backward subtests; 9-WAIS-III letter-number sequencing subtest; 10-WAIS-III vocabulary subtest that was used as measure of premorbid intelligence quotient (IQ); 11-Stroop Test; 12-letter (FAS) and semantic (animal) fluency tests; 14-Eyes Task; 15-Continuous Performance Test (CPT).

SUMMARY:
Cognitive enhancement is a primary goal in treating individuals with schizophrenia. Cognitive deficits are already present at the first break of the illness, seem to remain stable during early phases and noticeably influence daily functioning. Differences among antipsychotics in terms of cognitive effectiveness have turned out to be a topic of increasing research interest. The initially postulated superior neurocognitive effectiveness of second-generation antipsychotics (SGAs) compared to first-generation antipsychotics (FGAs) is currently under debate. Long-term studies would be of great value to evaluate the differential benefits exerted by antipsychotic drugs on cognitive performance. The aim of this study is to investigate the cognitive effects of aripiprazole, quetiapine and ziprasidone in first-episode psychosis at 1 year.

DETAILED DESCRIPTION:
Study setting and financial support: data for the present investigation were obtained from an ongoing epidemiological and three-year longitudinal intervention program of first-episode psychosis (PAFIP) conducted at the outpatient clinic and the inpatient unit at the University Hospital Marqués de Valdecilla, Spain. Conforming to international standards for research ethics, this program was approved by the local institutional review board. Patients meeting inclusion criteria and their families provided written informed consent to be included in the PAFIP. The Mental Health Services of Cantabria provided funding for implementing the program. No pharmaceutical company supplied any financial support.

Study design: this is a prospective, randomized, flexible-dose, open-label study. Investigators used a simple randomization procedure: a computer-generated randomization list was drawn up by a statistician. Dose ranges were 5-30 mg/day Aripiprazole, 40-160 mg/day Ziprasidone and 100-600 mg/day Quetiapine. Rapid titration schedule (5-day), until optimal dose was reached, was as a rule used unless severe side effects occur. At the treating physician's discretion, the dose and type of antipsychotic medication could be changed based on clinical efficacy and the profile of side effects during the follow-up period. Antimuscarinic medication, Lormetazepam and Clonazepam were permitted for clinical reasons. No antimuscarinic agents were administered prophylactically. Antidepressants (Sertraline) and mood stabilizers (lithium) were permitted if clinically needed.

Clinical assessment: the severity scale of the Clinical Global Impression (CGI) scale, the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Positive symptoms (SAPS), the Scale for the Assessment of Negative symptoms (SANS), the Calgary Depression Scale for Schizophrenia (CDSS) and the Young Mania Rating Scale (YMRS) were used to evaluate symptomatology. To assess general adverse event experiences, the Scale of the Udvalg for Kliniske Undersogelser (UKU), the Simpson-Angus Rating Scale (SARS) and the Barnes Akathisia Scale (BAS) were used. The same trained psychiatrist (BC-F) completed all clinical assessments. These clinical data are described at AZQ2005 study.

Neuropsychological assessment. Cognitive functioning was assessed in patients at 2 points: baseline and 1 year after the initialization of antipsychotic treatment. The cognitive assessment at baseline was carried out at 12 weeks after recruitment because this time is considered optimal for patients' stabilization. The evaluation required approximately 2 h and was carried out in the same day by the same neuropsychologist (R.A.-A and E.G.-R). The neuropsychological battery comprises 9 cognitive domains: information processing speed, motor dexterity, working memory, verbal learning, visuospatial abilities, delayed memory, attention, executive function and theory of mind.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP II) from October 2005 to January 2011.
* Experiencing their first episode of psychosis (First Episode of Psychosis is defined as that psychopathological state in which for the first time and regardless of its duration, the patient has enough severe psychotic symptoms to allow a diagnosis of psychosis, having received no specific psychiatric treatment for him).
* Living in the catchment area (Cantabria).
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for brief psychotic disorder, schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury with loss of consciousness.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Global cognitive index | 1 year
  In order to calculate a measure of Global Cognitive Functioning (GCF) raw cognitive scores were reversed when appropriate before standardization so they all have the same direction (the higher, the better). According to previous methodology, the GCF was calculated as T-scores, with raw scores of a healthy comparison sample. T scores were converted to deficit scores that reflect presence and severity of cognitive impairment. Deficit scores on all tests were then "averaged" to create the GCF score.

SECONDARY OUTCOMES:
Change in information processing speed | 1 year
  Measured by Wechsler Adult Intelligence Scale (WAIS) - III digit symbol subtest (standard total score), Trail Making Test (TMT) trail A and Continuous Performance Test (CPT) reaction time.
Change in motor dexterity | 1 year
  Measured by Grooved Pegboard Test (time to complete with dominant hand).
Change in working memory | 1 year
  Measured by WAIS - III letter-number sequencing test (standard total score) and WAIS - III digits forward (standard total score).
Change in verbal learning | 1 year
  Measured by the Rey Auditory Verbal Learning Test (RAVLT) (trials 1-5).
Change in visuospatial abilities | 1 year
  Measured by the Rey Complex Figure (RCF) (copy figure).
Change in delayed memory | 1 year
  Measured by RAVLT (list recall and list recognition discrimination subscore) and RCF (delayed recall).
Change in attention | 1 year
  Measured by CPT (discrimination subscores).
Change in executive function | 1 year
  Measured by TMT trail B, Stroop Test (color-word), the Zoo Map Test (first and second conditions), the Tower of London Test (ToL) (total correct and total moves score) and letter (FAS) and semantic (animal) fluency tests.
Change in theory of mind | 1 year
  Measured by Eyes Task (total correct score).

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Santander, Spain.
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brouwer RM, Klein M, Grasby KL, Schnack HG, Jahanshad N, Teeuw J, Thomopoulos SI, Sprooten E, Franz CE, Gogtay N, Kremen WS, Panizzon MS, Olde Loohuis LM, Whelan CD, Aghajani M, Alloza C, Alnaes D, Artiges E, Ayesa-Arriola R, Barker GJ, Bastin ME, Blok E, Boen E, Breukelaar IA, Bright JK, Buimer EEL, Bulow R, Cannon DM, Ciufolini S, Crossley NA, Damatac CG, Dazzan P, de Mol CL, de Zwarte SMC, Desrivieres S, Diaz-Caneja CM, Doan NT, Dohm K, Frohner JH, Goltermann J, Grigis A, Grotegerd D, Han LKM, Harris MA, Hartman CA, Heany SJ, Heindel W, Heslenfeld DJ, Hohmann S, Ittermann B, Jansen PR, Janssen J, Jia T, Jiang J, Jockwitz C, Karali T, Keeser D, Koevoets MGJC, Lenroot RK, Malchow B, Mandl RCW, Medel V, Meinert S, Morgan CA, Muhleisen TW, Nabulsi L, Opel N, de la Foz VO, Overs BJ, Paillere Martinot ML, Redlich R, Marques TR, Repple J, Roberts G, Roshchupkin GV, Setiaman N, Shumskaya E, Stein F, Sudre G, Takahashi S, Thalamuthu A, Tordesillas-Gutierrez D, van der Lugt A, van Haren NEM, Wardlaw JM, Wen W, Westeneng HJ, Wittfeld K, Zhu AH, Zugman A, Armstrong NJ, Bonfiglio G, Bralten J, Dalvie S, Davies G, Di Forti M, Ding L, Donohoe G, Forstner AJ, Gonzalez-Penas J, Guimaraes JPOFT, Homuth G, Hottenga JJ, Knol MJ, Kwok JBJ, Le Hellard S, Mather KA, Milaneschi Y, Morris DW, Nothen MM, Papiol S, Rietschel M, Santoro ML, Steen VM, Stein JL, Streit F, Tankard RM, Teumer A, van 't Ent D, van der Meer D, van Eijk KR, Vassos E, Vazquez-Bourgon J, Witt SH; IMAGEN Consortium; Adams HHH, Agartz I, Ames D, Amunts K, Andreassen OA, Arango C, Banaschewski T, Baune BT, Belangero SI, Bokde ALW, Boomsma DI, Bressan RA, Brodaty H, Buitelaar JK, Cahn W, Caspers S, Cichon S, Crespo-Facorro B, Cox SR, Dannlowski U, Elvsashagen T, Espeseth T, Falkai PG, Fisher SE, Flor H, Fullerton JM, Garavan H, Gowland PA, Grabe HJ, Hahn T, Heinz A, Hillegers M, Hoare J, Hoekstra PJ, Ikram MA, Jackowski AP, Jansen A, Jonsson EG, Kahn RS, Kircher T, Korgaonkar MS, Krug A, Lemaitre H, Malt UF, Martinot JL, McDonald C, Mitchell PB, Muetzel RL, Murray RM, Nees F, Nenadic I, Oosterlaan J, Ophoff RA, Pan PM, Penninx BWJH, Poustka L, Sachdev PS, Salum GA, Schofield PR, Schumann G, Shaw P, Sim K, Smolka MN, Stein DJ, Trollor JN, van den Berg LH, Veldink JH, Walter H, Westlye LT, Whelan R, White T, Wright MJ, Medland SE, Franke B, Thompson PM, Hulshoff Pol HE. Genetic variants associated with longitudinal changes in brain structure across the lifespan. Nat Neurosci. 2022 Apr;25(4):421-432. doi: 10.1038/s41593-022-01042-4. Epub 2022 Apr 5. PMID 35383335
- [Derived] Delgado-Alvarado M, Tordesillas-Gutierrez D, Ayesa-Arriola R, Canal M, de la Foz VO, Labad J, Crespo-Facorro B. Plasma prolactin levels are associated with the severity of illness in drug-naive first-episode psychosis female patients. Arch Womens Ment Health. 2019 Jun;22(3):367-373. doi: 10.1007/s00737-018-0899-x. Epub 2018 Aug 10. PMID 30097769
- [Derived] Tordesillas-Gutierrez D, Ayesa-Arriola R, Delgado-Alvarado M, Robinson JL, Lopez-Morinigo J, Pujol J, Dominguez-Ballesteros ME, David AS, Crespo-Facorro B. The right occipital lobe and poor insight in first-episode psychosis. PLoS One. 2018 Jun 1;13(6):e0197715. doi: 10.1371/journal.pone.0197715. eCollection 2018. PMID 29856773
- [Derived] Ayesa-Arriola R, Setien-Suero E, Neergaard KD, Belzunces AA, Contreras F, van Haren NEM, Crespo-Facorro B. Premorbid IQ subgroups in first episode non affective psychosis patients: Long-term sex differences in function and neurocognition. Schizophr Res. 2018 Jul;197:370-377. doi: 10.1016/j.schres.2017.12.006. Epub 2017 Dec 21. PMID 29275855